CLINICAL TRIAL: NCT00685360
Title: A Multi Center, Randomized, Double-blind, Placebo-controlled Phase 2 Trial to Evaluate the Safety, Efficacy and Pharmacokinetics of Multiple Doses of OPC 67683 in Patients With Pulmonary Sputum Culture-Positive, Multidrug-resistant Tuberculosis
Brief Title: A Trial to Evaluate OPC 67683 in Participants With Pulmonary Sputum Culture-positive, Multidrug-resistant Tuberculosis (TB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 242-07-204; 2007-005229-31 (EudraCT Number)
Record Dates: First submitted 2008-05-20; First posted 2008-05-28 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Multidrug Resistant; Extensively Drug-Resistant Tuberculosis
Keywords: Tuberculosis; Pulmonary; Multidrug resistant; Antitubercular Agents; OPC 67683
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis | interventions — OPC-67683

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Delamanid 100 mg BID + OBR (Experimental): Participants received delamanid 100 milligrams (mg) (two 50 mg tablets), orally, BID with two matching placebo tablets plus optimized background regimen (OBR) for 56 consecutive days (from Day 1 to Day 56).
  Participants were administered OBR as directed by the given investigator based on World Health Organization (WHO) guidelines and clinical judgment, in conjunction with national TB program guidelines in each country.
  Interventions: Drug: Delamanid; Drug: Optimized Background Regimen (OBR); Drug: Placebo
- Delamanid 200 mg BID + OBR (Experimental): Participants received delamanid 200 mg (four 50 mg tablets), orally, BID plus OBR for 56 consecutive days (from Day 1 to Day 56).
  Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment, in conjunction with national TB program guidelines in each country.
  Interventions: Drug: Delamanid; Drug: Optimized Background Regimen (OBR)
- Placebo + OBR (Placebo Comparator): Participants received four placebo tablets matching 50-mg tablets of delamanid, orally, BID plus OBR for 56 consecutive days (from Day 1 to Day 56).
  Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment, in conjunction with national TB program guidelines in each country.
  Interventions: Drug: Optimized Background Regimen (OBR); Drug: Placebo

INTERVENTIONS:
Drug: Delamanid — Delamanid was administered orally twice daily as 50-mg tablets under fed conditions in the morning and evening.
  Other Names: OPC-67683
  Arms: Delamanid 100 mg BID + OBR; Delamanid 200 mg BID + OBR
Drug: Optimized Background Regimen (OBR) — Selection and administration of the treatment medications (i.e., OBRs) was based on World Health Organization (WHO's) Guidelines for the programmatic management of drug-resistant TB, in conjunction with national TB program guidelines in each country.
  Study Investigator could change OBR for a participant based on participant's tolerability and drug susceptibility testing (DST) results.
Drug: Placebo — Placebo tablets matching 50-mg tablets of delamanid
  Arms: Delamanid 100 mg BID + OBR; Placebo + OBR

SUMMARY:
This is a clinical trial to evaluate the safety and efficacy of OPC-67683 in the treatment of multidrug resistant tuberculosis (MDR TB) for 56 days. In addition to an optimized background regimen (OBR), participants will be randomized to receive:

* 100 mg OPC-67683 twice daily (BID)
* 200 mg OPC-67683 BID
* Placebo BID

After 56 days participants will complete their optimized background regimen (OBR).

DETAILED DESCRIPTION:
This is a multi center, randomized, double-blinded, stratified, placebo-controlled clinical trial in three parallel groups. Participants will be randomized to one of the following three treatment groups:

* OBR plus 100 mg OPC-67683 BID
* OBR plus 200 mg OPC-67683 BID
* OBR plus placebo BID

The three treatment groups will comprise approximately 140 participants each (male or female). The trial will consist of the following periods:

* Pre-treatment Period (Visits 1 to 3 [Day -9 to Day -1])
* Treatment Period (Visits 4 to 59 [Days 1 to 56])
* Post-treatment Period (Visits 60 to 64 [Days 57 to 84])

Enrolled participants (those accepted into the screening period of the trial who signed an informed consent form) will be stratified at randomization by extent of pulmonary TB; an equal number of participants with and without cavities visible in the lung fields on baseline chest radiograph will be allocated to each treatment group. A total of approximately 430 male or female participants aged 18 to 64 years, inclusive, with pulmonary, sputum culture-positive MDR TB (TB caused by Mycobacterium tuberculosis strains resistant to at least isoniazid and rifampicin) or with sputum smears positive for acid fast bacilli (AFB) and a positive rapid test for rifampicin resistance on direct sputum within 60 days prior to the expected date of enrollment. Participants with positive AFB smears and a positive rapid rifampicin resistance test will be enrolled as presumptively culture positive and withdrawn as ineligible if they are confirmed to not have sputum culture positive MDR TB.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures
* Male and female participants aged between 18 and 64 years, inclusive.
* Either mycobacterial culture of sputum positive for growth of Mycobacterium tuberculosis or sputum smear positive for acid fast bacilli within 60 days prior to the expected date of enrollment.
* Participant with TB caused by isolates of Mycobacterium tuberculosis complex confirmed to be resistant to treatment with isoniazid and rifampicin, or with positive rapid test for rifampicin resistance on direct sputum positive for acid fast bacilli within 60 days prior to the expected date of enrollment.
* Findings on chest radiograph consistent with TB.
* Able to produce sputum for mycobacterial culture.
* Female participants of childbearing potential must have a negative urine pregnancy test and agree to use a highly effective method of birth control (for example, two of the following precautions: tubal ligation, vaginal diaphragm, intrauterine device, oral contraceptives, contraceptive implant, combined hormonal patch, combined injectable contraceptive or depot-medroxyprogesterone acetate) throughout the participation in the trial and for 22 weeks after last dose (to cover duration of ovulation).
* Male participants must agree to use an adequate method of contraception (double barrier) throughout the participation in the trial and for 30 weeks after last dose (to cover duration of spermatogenesis).

Exclusion Criteria:

* A history of allergy to any nitro-imidazoles or nitro-imidazole derivates at any time.
* Use of the medications including: use of amiodarone at any time during the previous 12 months, use of other anti-arrhythmics for the previous 30 days, and use of certain other medications, including certain anti-depressants, anti-histamines, and macrolides, for the previous 14 days.
* Any current serious concomitant conditions or renal impairment characterized by serum creatinine levels ≥265 micromol/L or hepatic impairment characterized by alanine transaminase (ALT) and/or aspartate transferase (AST) levels 3 times the upper limit of the laboratory reference range.
* Current clinically relevant changes in the electrocardiogram (ECG) such as any atrioventricular (AV) block, prolongation of the QRS complex over 120 milliseconds (in both male and female participants), or of either the QT interval corrected by Fridericia's formula (QTcF) or QT interval corrected by Bazett's formula (QTcB) interval over 430 milliseconds in male participants and 450 milliseconds in female participants.
* Current clinically relevant cardiovascular disorder such as heart failure, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia or status after myocardial infarction.
* For participants with human immunodeficiency virus (HIV) infection, cluster of differentiation 4 helper/inducer T cell[s] (CD4) cell count < 350/mm3 or on treatment with anti-retroviral medication for HIV infection.
* Karnofsky score < 60%.
* Any diseases or conditions in which the use of nitro-imidazoles or nitro-imidazole derivates is contra-indicated.
* Evidence of clinically significant metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied).
* Known or suspected alcohol abuse, that is, abuse sufficient enough to compromise the safety or cooperation of the participant in the opinion of the investigator.
* Administered an investigational medicinal product (IMP) within 1 month prior to Visit 1 (Screening [Days -9 to -3]).
* Pregnant, breast-feeding, or planning to conceive or father a child within the timeframe described in the informed consent form.
* Recent use of methadone, benzodiazepines, cocaine, amphetamine/metamphetamine, tetrahydrocannabinol, barbiturates, tricyclic antidepressants, and opiates as determined by a urine drug screen unless evidence is provided that the positive drug screen is the result of authorized medications products prescribed by a physician for a non-abuse-related indication.
* Any disorder that in the judgment of the investigator makes the participant not a good candidate for the trial or may prevent the participant from reliably participating in the entire course of the trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 481 (Actual)
Dates: Start 2008-05-08 (Actual); Primary Completion 2010-06-11 (Actual); Study Completion 2010-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (17):
- University of Texas Health Center at Tyler / Heartland National TB Center / Texas Center for Infectious Disease, San Antonio, Texas, United States
- China (2):
  - Beijing Chest Hospital, Beijing
  - Shanghai Pulmonary Hospital, Shanghai
- Abbassia Chest Hospital, Cairo, Egypt
- Estonia (2):
  - North Estonian Medical Centre Foundation, Tallinn
  - Tartu University Lung Hospital, Tartu
- Japan (2):
  - Kinki Chuo Chest Hospital, Osaka
  - Fukujuji Hospital, Tokyo
- Clinic of Tuberculosis and Lung Diseases, Riga, Latvia
- Peru (3):
  - Hospital Nacional Daniel Alcides Carrión, Carrion
  - Hospital Nacional Sergio E. Bernales, Lima
  - Hospital Nacional Hipolito Unanue, Unánue
- Tropical Disease Foundation, Manila, Philippines
- South Korea (4):
  - Masan Medical Center, Changwon
  - National Masan Hospital, Masan
  - Younsei University Medical Center (YUMC), Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Gler MT, Skripconoka V, Sanchez-Garavito E, Xiao H, Cabrera-Rivero JL, Vargas-Vasquez DE, Gao M, Awad M, Park SK, Shim TS, Suh GY, Danilovits M, Ogata H, Kurve A, Chang J, Suzuki K, Tupasi T, Koh WJ, Seaworth B, Geiter LJ, Wells CD. Delamanid for multidrug-resistant pulmonary tuberculosis. N Engl J Med. 2012 Jun 7;366(23):2151-60. doi: 10.1056/NEJMoa1112433. PMID 22670901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 17 investigative sites in the Philippines, Latvia, Estonia, South Korea, Peru, China, Japan, Egypt, and the United States from 08 May 2008 to 11 June 2010.
Pre-assignment Details: Participants with pulmonary sputum culture-positive, multidrug-resistant tuberculosis were randomized in 1:1:1 ratio to 1 of the 3 groups to receive either optimized background regimen (OBR) + 100 milligrams (mg) BID delamanid or OBR + 200 mg BID delamanid or OBR + placebo.
Groups:
- Delamanid 100 mg BID + OBR: Participants received delamanid 100 mg (two 50 mg tablets), orally, twice daily (BID) with two matching placebo tablets plus OBR for 56 consecutive days (from Day 1 to Day 56).
  Participants were administered OBR as directed by the given investigator based on World Health Organization (WHO) guidelines and clinical judgment, in conjunction with national TB program guidelines in each country.
Period: Overall Study
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Started | 161 | 160 | 160
Modified Intent-to-Treat (MITT) (MITT Population included all participants who had sputum cultures positive for multidrug resistant tuberculosis (MDR TB) at baseline (Day -1 and/or Day 1) using the mycobacteria growth indicator tube (MGIT) system.) | 141 | 136 | 125
MITT (Solid Culture) (MITT (Solid Culture) Population included all participants who had sputum cultures positive for MDR TB at baseline (Day -1 and/or Day 1) using solid culture medium.) | 119 | 115 | 113
Completed | 143 | 146 | 145
Not Completed | 18 | 14 | 15
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Adverse Event | 4 | 6 | 4
Not completed — Subject Met (Protocol Specified) Withdrawal Criteria | 1 | 0 | 2
Not completed — Subject was Withdrawn From Participation by the Investigator | 0 | 4 | 1
Not completed — Subject Withdrew Consent to Participate | 13 | 2 | 5
Not completed — Protocol Deviation | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population included all randomized participants who received any amount of investigational medicinal product (IMP), regardless of any protocol deviation or violation.
Groups:
- Delamanid 100 mg BID + OBR: Participants received delamanid 100 mg (two 50 mg tablets), orally, BID with two matching placebo tablets plus OBR for 56 consecutive days (from Day 1 to Day 56).
  Participants were administered OBR as directed by the given investigator based on WHO guidelines and clinical judgment, in conjunction with national TB program guidelines in each country.
- Total: Total of all reporting groups
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR | Total
Number analyzed (Participants) | 161 | 160 | 160 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.1) | 35.4 (12.0) | 36.1 (11.4) | 36.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 52 | 49 | 157
  Male | 105 | 108 | 111 | 324
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 44 | 47 | 133
  Not Hispanic or Latino | 118 | 116 | 113 | 347
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 38 | 31 | 26 | 95
  Race: Black or African American | 0 | 1 | 0 | 1
  Race: Asian | 82 | 87 | 88 | 257
  Race: Other | 41 | 41 | 46 | 128

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Sputum Culture Conversion (SCC) Using the Mycobacteria Growth Indicator Tube (MGIT) System
Description: Sputum culture conversion was defined to occur at the time of the collection of a sputum specimen with mycobacterial culture negative for growth of Mycobacterium tuberculosis (MTB) followed by at least one additional sputum specimen with mycobacterial culture negative for growth at least 27 days after the first negative specimen and not followed by any sputum specimens positive for growth in the MGIT system at any point during the remainder of the 84-day trial after the first negative culture.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 84)
Population: Modified Intent-to-Treat (MITT) Population included all participants who had sputum cultures positive for multidrug resistant tuberculosis (MDR TB) at baseline (Day -1 and/or Day 1) using the MGIT system.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 141 | 136 | 125
percentage of participants | 45.4 | 41.9 | 29.6
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0083, Cochran-Mantel-Haenszel; P-value was derived using Cochran-Mantel-Haenszel (CMH) test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.534, 95% CI 2-sided [1.107 to 2.124]
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0393, Cochran-Mantel-Haenszel — P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.416, 95% CI 2-sided [1.012 to 1.980]

2. Primary Outcome: Tmax 1 and 2: Time to Maximal Peak Concentration (Tmax) for Delamanid Following First and Second Daily Dose
Description: Time to maximum (peak) plasma concentration following the first daily dose (Cmax1) was reported as tmax1 and time to maximum (peak) plasma concentration following the second daily dose (Cmax2) was reported as tmax2. Data for Tmax up to Day 56 was collected on Days 1, 14, 28 and 56.
Time Frame: Pre-dose, 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: All randomized participants who received at least one dose of study medication. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
hours
  Day 1: tmax1: number analyzed (Participants) | 159 | 159
  Day 1: tmax1 | 4.00 [1.85 to 10.0] | 4.00 [2.00 to 10.0]
  Day 1: tmax2: number analyzed (Participants) | 159 | 159
  Day 1: tmax2 | 14.0 [11.7 to 24.0] | 14.0 [11.9 to 24.0]
  Day 14: tmax1: number analyzed (Participants) | 150 | 153
  Day 14: tmax1 | 3.02 [0.00 to 10.0] | 3.00 [0.00 to 10.0]
  Day 14: tmax2: number analyzed (Participants) | 150 | 153
  Day 14: tmax2 | 14.0 [11.9 to 24.0] | 14.0 [12.0 to 24.0]
  Day 28: tmax1: number analyzed (Participants) | 145 | 150
  Day 28: tmax1 | 3.02 [0.00 to 10.0] | 3.00 [0.00 to 10.0]
  Day 28: tmax2: number analyzed (Participants) | 145 | 150
  Day 28: tmax2 | 14.0 [12.0 to 24.0] | 14.0 [12.0 to 24.0]
  Day 56: tmax1: number analyzed (Participants) | 144 | 145
  Day 56: tmax1 | 3.02 [0.00 to 9.97] | 3.02 [0.00 to 10.0]
  Day 56: tmax2: number analyzed (Participants) | 144 | 145
  Day 56: tmax2 | 14.0 [12.0 to 24.0] | 14.0 [12.0 to 24.0]

3. Primary Outcome: Cmax 1 and 2: Maximal Peak Concentration (Cmax) for Delamanid Following First and Second Daily Dose
Description: Maximum (peak) plasma concentration following the first daily dose was reported as Cmax1 and maximum (peak) plasma concentration following the second daily dose was reported as Cmax2. Data for Cmax up to Day 56 was collected on Days 1, 14, 28 and 56.
Time Frame: Pre-dose, 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mL
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
nanograms (ng)/mL
  Day 1: Cmax1: number analyzed (Participants) | 159 | 159
  Day 1: Cmax1 | 135 (54.9) | 187 (74.3)
  Day 1: Cmax2: number analyzed (Participants) | 159 | 159
  Day 1: Cmax2 | 151 (60.4) | 228 (91.5)
  Day 14: Cmax1: number analyzed (Participants) | 150 | 153
  Day 14: Cmax1 | 369 (137) | 547 (200)
  Day 14: Cmax2: number analyzed (Participants) | 150 | 153
  Day 14: Cmax2 | 361 (127) | 513 (178)
  Day 28: Cmax1: number analyzed (Participants) | 145 | 150
  Day 28: Cmax1 | 404 (144) | 599 (222)
  Day 28: Cmax2: number analyzed (Participants) | 145 | 150
  Day 28: Cmax2 | 381 (128) | 560 (196)
  Day 56: Cmax1: number analyzed (Participants) | 144 | 145
  Day 56: Cmax1 | 414 (165) | 611 (217)
  Day 56: Cmax2: number analyzed (Participants) | 144 | 145
  Day 56: Cmax2 | 400 (162) | 588 (213)

4. Primary Outcome: Area Under the Plasma Concentration Curve From 0 to 24 Hours (AUC0-24h) for Delamanid
Description: Data for AUC0-24h up to Day 56 was collected on Days 1, 14, 28 and 56.
Time Frame: Pre-dose, 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours*nanograms (h*ng)/mL
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
hours*nanograms (h*ng)/mL
  Day 1: AUC0-24h: number analyzed (Participants) | 159 | 159
  Day 1: AUC0-24h | 2441 (880) | 3598 (1312)
  Day 14: AUC0-24h: number analyzed (Participants) | 150 | 153
  Day 14: AUC0-24h | 7234 (2346) | 10490 (3377)
  Day 28: AUC0-24h: number analyzed (Participants) | 145 | 150
  Day 28: AUC0-24h | 7700 (2322) | 11251 (3626)
  Day 56: AUC0-24h: number analyzed (Participants) | 144 | 145
  Day 56: AUC0-24h | 7925 (2973) | 11837 (3975)

5. Primary Outcome: Accumulation Ratio for Cmax (Rac[Cmax]) for Delamanid
Description: Data for Rac (Cmax) up to Day 56 was collected on Days 14, 28 and 56. Rac (Cmax) on Days 14, 28 or 56 compared to Cmax on Day 1 was computed.
Time Frame: Pre-dose, 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
ratio
  Day 14: Rac Cmax1: number analyzed (Participants) | 150 | 152
  Day 14: Rac Cmax1 | 3.05 (1.28) | 4.74 (19.5)
  Day 14: Rac Cmax2: number analyzed (Participants) | 150 | 152
  Day 14: Rac Cmax2 | 2.65 (1.11) | 2.43 (0.870)
  Day 28: Rac Cmax1: number analyzed (Participants) | 145 | 149
  Day 28: Rac Cmax1 | 3.35 (1.63) | 4.94 (18.0)
  Day 28: Rac Cmax2: number analyzed (Participants) | 145 | 149
  Day 28: Rac Cmax2 | 2.85 (1.65) | 2.65 (1.01)
  Day 56: Rac Cmax1: number analyzed (Participants) | 144 | 144
  Day 56: Rac Cmax1 | 3.37 (1.46) | 5.09 (18.0)
  Day 56: Rac Cmax2: number analyzed (Participants) | 144 | 144
  Day 56: Rac Cmax2 | 2.92 (1.43) | 2.81 (1.19)

6. Primary Outcome: Accumulation Ratio for AUC From Time 0 to 24 Hours (Rac[AUC0-24h]) for Delamanid
Description: Data for Rac (AUC) up to Day 56 was collected on Days 14, 28 and 56. Rac (AUC) on Days 14, 28 or 56 compared to AUC0-24h on Day 1 was computed.
Time Frame: Pre-dose, 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
ratio
  Day 14: Rac AUC0-24h: number analyzed (Participants) | 150 | 152
  Day 14: Rac AUC0-24h | 3.14 (0.965) | 3.13 (1.06)
  Day 28: Rac AUC0-24h: number analyzed (Participants) | 145 | 149
  Day 28: Rac AUC0-24h | 3.35 (1.24) | 3.33 (1.12)
  Day 56: Rac AUC0-24h: number analyzed (Participants) | 144 | 144
  Day 56: Rac AUC0-24h | 3.41 (1.19) | 3.52 (1.38)

7. Primary Outcome: Time to Maximal Peak Concentration (Tmax) for Delamanid Metabolite (DM)-6704, DM-6705, DM-6706, DM-6717, DM-6718, DM-6720, DM-6721, and DM-6722
Description: Data for Tmax up to Day 56 was collected on Days 1, 14, 28 and 56.
Time Frame: 0 hours (morning pre-dose), 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: All randomized participants who received at least one dose of study medication. Number analyzed is the number of participants with data available for analysis at the given time point for the specified category.
Measure: Median (Full Range); unit: hours
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
hours
  All Metabolites: Tmax at Day 1 | NA [NA to NA] — Data is not available as the concentration of metabolites was below the level of detection on Day 1. | NA [NA to NA] — Data is not available as the concentration of metabolites was below the level of detection on Day 1.
  DM-6704: Tmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6704: Tmax at Day 14 | 13.0 [0.00 to 24.0] | 13.0 [0.00 to 24.0]
  DM-6704: Tmax at Day 28: number analyzed (Participants) | 145 | 150
  DM-6704: Tmax at Day 28 | 3.97 [0.00 to 24.0] | 3.99 [0.00 to 24.0]
  DM-6704: Tmax at Day 56: number analyzed (Participants) | 143 | 145
  DM-6704: Tmax at Day 56 | 3.97 [0.00 to 24.0] | 4.00 [0.00 to 24.0]
  DM-6705: Tmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6705: Tmax at Day 14 | 12.0 [0.00 to 24.0] | 9.97 [0.00 to 24.0]
  DM-6705: Tmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6705: Tmax at Day 28 | 9.97 [0.00 to 24.0] | 9.97 [0.00 to 24.0]
  DM-6705: Tmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6705: Tmax at Day 56 | 9.97 [0.00 to 24.0] | 12.0 [0.00 to 24.0]
  DM-6706: Tmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6706: Tmax at Day 14 | 14.0 [0.00 to 24.0] | 12.0 [0.00 to 24.0]
  DM-6706: Tmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6706: Tmax at Day 28 | 3.01 [0.00 to 24.0] | 4.00 [0.00 to 24.0]
  DM-6706: Tmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6706: Tmax at Day 56 | 3.03 [0.00 to 24.0] | 4.00 [0.00 to 24.0]
  DM-6717: Tmax at Day 14: number analyzed (Participants) | 147 | 153
  DM-6717: Tmax at Day 14 | 24.0 [0.00 to 24.0] | 24.0 [0.00 to 24.0]
  DM-6717: Tmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6717: Tmax at Day 28 | 9.99 [0.00 to 24.0] | 13.0 [0.00 to 24.0]
  DM-6717: Tmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6717: Tmax at Day 56 | 9.97 [0.00 to 24.0] | 9.99 [0.00 to 24.0]
  DM-6718: Tmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6718: Tmax at Day 14 | 24.0 [0.00 to 24.0] | 24.0 [0.00 to 24.0]
  DM-6718: Tmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6718: Tmax at Day 28 | 10.0 [0.00 to 24.0] | 12.9 [0.00 to 24.0]
  DM-6718: Tmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6718: Tmax at Day 56 | 9.96 [0.00 to 24.0] | 9.97 [0.00 to 24.0]
  DM-6720: Tmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6720: Tmax at Day 14 | 11.0 [0.00 to 24.0] | 10.0 [0.00 to 24.0]
  DM-6720: Tmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6720: Tmax at Day 28 | 9.97 [0.00 to 24.0] | 9.97 [0.00 to 24.0]
  DM-6720: Tmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6720: Tmax at Day 56 | 9.97 [0.00 to 24.0] | 9.97 [0.00 to 24.0]
  DM-6721: Tmax at Day 14: number analyzed (Participants) | 130 | 148
  DM-6721: Tmax at Day 14 | 13.0 [0.00 to 24.0] | 10.0 [0.00 to 24.0]
  DM-6721: Tmax at Day 28: number analyzed (Participants) | 144 | 149
  DM-6721: Tmax at Day 28 | 4.02 [0.00 to 24.0] | 4.00 [0.00 to 24.0]
  DM-6721: Tmax at Day 56: number analyzed (Participants) | 139 | 144
  DM-6721: Tmax at Day 56 | 4.02 [0.00 to 24.0] | 9.97 [0.00 to 24.0]
  DM-6722: Tmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6722: Tmax at Day 14 | 13.0 [0.00 to 24.0] | 9.98 [0.00 to 24.0]
  DM-6722: Tmax at Day 28: number analyzed (Participants) | 145 | 150
  DM-6722: Tmax at Day 28 | 3.00 [0.00 to 24.0] | 4.00 [0.00 to 24.0]
  DM-6722: Tmax at Day 56: number analyzed (Participants) | 143 | 145
  DM-6722: Tmax at Day 56 | 4.00 [0.00 to 24.0] | 4.00 [0.00 to 24.0]

8. Primary Outcome: Maximal Peak Concentration (Cmax) for DM-6704, DM-6705, DM-6706, DM-6717, DM-6718, DM-6720, DM-6721, and DM-6722
Description: Data for Cmax up to Day 56 was collected on Days 1, 14, 28 and 56.
Time Frame: 0 hours (morning pre-dose), 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
ng/mL
  All Metabolites: Cmax at Day 1 | NA (NA) — Data is not available as the concentration of metabolites was below the level of detection on Day 1. | NA (NA) — Data is not available as the concentration of metabolites was below the level of detection on Day 1.
  DM-6704: Cmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6704: Cmax at Day 14 | 40.9 (29.9) | 57.1 (40.7)
  DM-6704: Cmax at Day 28: number analyzed (Participants) | 145 | 150
  DM-6704: Cmax at Day 28 | 48.9 (31.4) | 78.3 (53.0)
  DM-6704: Cmax at Day 56: number analyzed (Participants) | 143 | 145
  DM-6704: Cmax at Day 56 | 60.6 (37.7) | 90.3 (58.5)
  DM-6705: Cmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6705: Cmax at Day 14 | 78.3 (35.1) | 124 (57.8)
  DM-6705: Cmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6705: Cmax at Day 28 | 121 (57.4) | 187 (78.5)
  DM-6705: Cmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6705: Cmax at Day 56 | 151 (67.3) | 233 (94.5)
  DM-6706: Cmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6706: Cmax at Day 14 | 32.5 (15.9) | 46.5 (24.2)
  DM-6706: Cmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6706: Cmax at Day 28 | 47.1 (22.1) | 69.9 (32.0)
  DM-6706: Cmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6706: Cmax at Day 56 | 59.2 (30.5) | 84.3 (41.5)
  DM-6717: Cmax at Day 14: number analyzed (Participants) | 147 | 153
  DM-6717: Cmax at Day 14 | 5.44 (4.04) | 7.61 (4.51)
  DM-6717: Cmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6717: Cmax at Day 28 | 16.9 (11.7) | 25.5 (17.0)
  DM-6717: Cmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6717: Cmax at Day 56 | 34.7 (20.5) | 53.4 (30.3)
  DM-6718: Cmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6718: Cmax at Day 14 | 26.6 (20.2) | 32.6 (17.1)
  DM-6718: Cmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6718: Cmax at Day 28 | 66.5 (34.9) | 84.9 (34.5)
  DM-6718: Cmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6718: Cmax at Day 56 | 107 (46.6) | 138 (47.9)
  DM-6720: Cmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6720: Cmax at Day 14 | 19.5 (11.7) | 26.5 (11.6)
  DM-6720: Cmax at Day 28: number analyzed (Participants) | 146 | 150
  DM-6720: Cmax at Day 28 | 39.4 (17.1) | 53.6 (18.7)
  DM-6720: Cmax at Day 56: number analyzed (Participants) | 144 | 146
  DM-6720: Cmax at Day 56 | 57.4 (22.6) | 79.3 (26.3)
  DM-6721: Cmax at Day 14: number analyzed (Participants) | 130 | 148
  DM-6721: Cmax at Day 14 | 3.19 (2.26) | 4.38 (3.35)
  DM-6721: Cmax at Day 28: number analyzed (Participants) | 144 | 149
  DM-6721: Cmax at Day 28 | 4.95 (4.37) | 7.74 (6.37)
  DM-6721: Cmax at Day 56: number analyzed (Participants) | 139 | 144
  DM-6721: Cmax at Day 56 | 6.38 (5.65) | 9.92 (7.04)
  DM-6722: Cmax at Day 14: number analyzed (Participants) | 150 | 153
  DM-6722: Cmax at Day 14 | 23.1 (22.1) | 33.4 (27.3)
  DM-6722: Cmax at Day 28: number analyzed (Participants) | 145 | 150
  DM-6722: Cmax at Day 28 | 31.2 (31.8) | 48.5 (41.3)
  DM-6722: Cmax at Day 56: number analyzed (Participants) | 143 | 145
  DM-6722: Cmax at Day 56 | 33.3 (23.0) | 56.1 (39.7)

9. Primary Outcome: Area Under the Plasma Concentration Curve From 0 to 24 Hours (AUC0-24h) for DM-6704, DM-6705, DM-6706, DM-6717, DM-6718, DM-6720, DM-6721, and DM-6722
Description: Data for AUC0-24h up to Day 56 was collected on Days 1, 14, 28 and 56.
Time Frame: 0 hours (morning pre-dose), 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
h*ng/mL
  All Metabolites: AUC0-24h at Day 1 | NA (NA) — Data is not available as the concentration of metabolites was below the level of detection on Day 1. | NA (NA) — Data is not available as the concentration of metabolites was below the level of detection on Day 1.
  DM-6704: AUC0-24h at Day 14: number analyzed (Participants) | 150 | 153
  DM-6704: AUC0-24h at Day 14 | 848 (647) | 1192 (859)
  DM-6704: AUC0-24h at Day 28: number analyzed (Participants) | 145 | 150
  DM-6704: AUC0-24h at Day 28 | 1022 (679) | 1610 (1097)
  DM-6704: AUC0-24h at Day 56: number analyzed (Participants) | 143 | 145
  DM-6704: AUC0-24h at Day 56 | 1251 (766) | 1902 (1252)
  DM-6705: AUC0-24h at Day 14: number analyzed (Participants) | 150 | 153
  DM-6705: AUC0-24h at Day 14 | 1597 (632) | 2485 (920)
  DM-6705: AUC0-24h at Day 28: number analyzed (Participants) | 146 | 150
  DM-6705: AUC0-24h at Day 28 | 2480 (1051) | 3857 (1486)
  DM-6705: AUC0-24h at Day 56: number analyzed (Participants) | 144 | 146
  DM-6705: AUC0-24h at Day 56 | 3125 (1397) | 4907 (1987)
  DM-6706: AUC0-24h at Day 14: number analyzed (Participants) | 150 | 153
  DM-6706: AUC0-24h at Day 14 | 685 (339) | 992 (525)
  DM-6706: AUC0-24h at Day 28: number analyzed (Participants) | 146 | 150
  DM-6706: AUC0-24h at Day 28 | 1004 (474) | 1475 (676)
  DM-6706: AUC0-24h at Day 56: number analyzed (Participants) | 144 | 146
  DM-6706: AUC0-24h at Day 56 | 1256 (643) | 1796 (870)
  DM-6717: AUC0-24h at Day 14: number analyzed (Participants) | 145 | 153
  DM-6717: AUC0-24h at Day 14 | 108 (81.9) | 153 (93.2)
  DM-6717: AUC0-24h at Day 28: number analyzed (Participants) | 146 | 150
  DM-6717: AUC0-24h at Day 28 | 349 (240) | 524 (342)
  DM-6717: AUC0-24h at Day 56: number analyzed (Participants) | 144 | 146
  DM-6717: AUC0-24h at Day 56 | 720 (436) | 1112 (623)
  DM-6718: AUC0-24h at Day 14: number analyzed (Participants) | 150 | 153
  DM-6718: AUC0-24h at Day 14 | 528 (360) | 687 (363)
  DM-6718: AUC0-24h at Day 28: number analyzed (Participants) | 146 | 150
  DM-6718: AUC0-24h at Day 28 | 1424 (757) | 1800 (726)
  DM-6718: AUC0-24h at Day 56: number analyzed (Participants) | 144 | 146
  DM-6718: AUC0-24h at Day 56 | 2285 (992) | 2954 (994)
  DM-6720: AUC0-24h at Day 14: number analyzed (Participants) | 150 | 153
  DM-6720: AUC0-24h at Day 14 | 396 (193) | 551 (222)
  DM-6720: AUC0-24h at Day 28: number analyzed (Participants) | 146 | 150
  DM-6720: AUC0-24h at Day 28 | 822 (353) | 1120 (368)
  DM-6720: AUC0-24h at Day 56: number analyzed (Participants) | 144 | 146
  DM-6720: AUC0-24h at Day 56 | 1206 (474) | 1668 (549)
  DM-6721: AUC0-24h at Day 14: number analyzed (Participants) | 128 | 146
  DM-6721: AUC0-24h at Day 14 | 65.4 (49.7) | 90.5 (68.7)
  DM-6721: AUC0-24h at Day 28: number analyzed (Participants) | 142 | 148
  DM-6721: AUC0-24h at Day 28 | 103 (92.9) | 161 (134)
  DM-6721: AUC0-24h at Day 56: number analyzed (Participants) | 139 | 144
  DM-6721: AUC0-24h at Day 56 | 132 (118) | 210 (154)
  DM-6722: AUC0-24h at Day 14: number analyzed (Participants) | 150 | 153
  DM-6722: AUC0-24h at Day 14 | 482 (475) | 707 (589)
  DM-6722: AUC0-24h at Day 28: number analyzed (Participants) | 145 | 150
  DM-6722: AUC0-24h at Day 28 | 655 (695) | 1013 (883)
  DM-6722: AUC0-24h at Day 56: number analyzed (Participants) | 143 | 145
  DM-6722: AUC0-24h at Day 56 | 699 (489) | 1191 (862)

10. Primary Outcome: Accumulation Ratio for Cmax (Rac[Cmax]) for DM-6704, DM-6705, DM-6706, DM-6717, DM-6718, DM-6720, DM-6721, and DM-6722
Description: Data for Rac (Cmax) up to Day 56 was to be collected on Days 1, 14, 28 and 56. Rac (Cmax) on Days 14, 28 or 56 compared to Cmax on Day 1 was to be computed. Due to limited measurable data on Day 1 for delamanid metabolites, pharmacokinetic (PK) analysis was not conducted on Day 1 data for delamanid metabolites, and data for Rac (Cmax) was not available.
Time Frame: 0 hours (morning pre-dose), 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: Due to limited measurable data as the metabolite concentration was below the level of detection on Day 1 for delamanid metabolites, PK analysis was not conducted on Day 1 data for delamanid metabolites, and data for Rac (Cmax) was not available.
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Accumulation Ratio for AUC (Rac[AUC]) for DM-6704, DM-6705, DM-6706, DM-6717, DM-6718, DM-6720, DM-6721, and DM-6722
Description: Data for Rac (AUC) up to Day 56 was to be collected on Days 1, 14, 28 and 56. Rac (AUC) on Days 14, 28 or 56 compared to AUC0-24h on Day 1 was to be computed. Due to limited measurable data on Day 1 for delamanid metabolites, PK analysis was not conducted on Day 1 data for delamanid metabolites, and data for Rac (AUC) was not available.
Time Frame: 0 hours (morning pre-dose), 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose up to Day 56
Population: Due to limited measurable data as the metabolite concentration was below the level of detection on Day 1 for delamanid metabolites, PK analysis was not conducted on Day 1 data for delamanid metabolites, and data for Rac (AUC) was not available.
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Elimination Half-life (t1/2) for DM-6704, DM-6705, DM-6706, DM-6717, DM-6718, DM-6720, DM-6721, and DM-6722
Time Frame: 0 hours (morning pre-dose), 2, 3, 4, 10 (pre-evening dose), 12, 13, 14 and 24 hours post-dose on Day 56
Population: All randomized participants who received at least one dose of study medication. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR
Number analyzed (Participants) | 161 | 160
hours
  t1/2 for DM-6704: number analyzed (Participants) | 116 | 127
  t1/2 for DM-6704 | 195 (115) | 191 (67.2)
  t1/2 for DM-6705: number analyzed (Participants) | 140 | 143
  t1/2 for DM-6705 | 231 (84.7) | 233 (87.9)
  t1/2 for DM-6706: number analyzed (Participants) | 137 | 141
  t1/2 for DM-6706 | 180 (43.1) | 184 (40.3)
  t1/2 for DM-6717: number analyzed (Participants) | 117 | 127
  t1/2 for DM-6717 | 265 (98.2) | 265 (115)
  t1/2 for DM-6718: number analyzed (Participants) | 102 | 88
  t1/2 for DM-6718 | 302 (132) | 305 (131)
  t1/2 for DM-6720: number analyzed (Participants) | 85 | 92
  t1/2 for DM-6720 | 394 (158) | 424 (192)
  t1/2 for DM-6721: number analyzed (Participants) | 18 | 31
  t1/2 for DM-6721 | 168 (49.7) | 153 (53.1)
  t1/2 for DM-6722: number analyzed (Participants) | 52 | 66
  t1/2 for DM-6722 | 134 (85.1) | 148 (60.3)

13. Secondary Outcome: Percentage of Participants Who Achieved Sputum Culture Conversion (SCC) Using Solid Culture Media
Description: A participant achieving SCC using solid culture media was defined as one with sputum culture negative for growth of MTB on Day 57, and (a) not followed by a positive culture at any point thereafter, and (b) confirmed by at least one additional negative sputum culture at Day 84.
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 84)
Population: MITT (Solid Culture) Population included all participants who had sputum cultures positive for MDR TB at baseline (Day -1 and/or Day 1) using solid culture medium.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 119 | 115 | 113
percentage of participants | 53.8 | 65.2 | 33.6
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.599, 95% CI 2-sided [1.175 to 2.177]
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Risk Ratio Mean = 1.939, 95% CI 2-sided [1.449 to 2.595]

14. Secondary Outcome: Change From Baseline in Time to Culture Positivity Using the MGIT System
Description: Mean change from baseline in time to culture positivity using the MGIT system was the value for "time to results" when a sputum culture result was positive (in days) using the MGIT system during the routine 42-day incubation period. A longer time to culture positivity represented a lower burden of MTB organisms present in the sputum. Baseline was defined as the average of Day -1 and Day 1 values, if the cultures on both days were positive; if only one culture was positive, the value for the positive culture was used as baseline.
Time Frame: Baseline, Day 84
Population: Last Observation Carried Forward(LOCF)Population:all randomized participants with positive sputum culture for MDR TB at baseline(pre-dose)by MGIT system and when sputum collection was not possible,a specimen was contaminated with other bacteria,or a result was missing due to a participant withdrawing from trial, the preceding non-missing result for that variable at a postbaseline visit was carried forward. Overall number analyzed=participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 140 | 135 | 123
days | 25.9 (1.0) | 26.0 (1.0) | 24.2 (1.1)
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.2419, ANCOVA; Pairwise comparison was derived from analysis of covariance(ANCOVA)model with factors of treatment, baseline cavitation status and covariate baseline
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.2239, ANCOVA; Pairwise comparison is derived from ANCOVA model with factors of treatment, baseline cavitation status and covariate baseline
Statistical Analysis 3: Comparison: Delamanid 100 mg BID + OBR vs Delamanid 200 mg BID + OBR; Test type: Superiority; p = 0.9544, ANCOVA; [statistical method as in outcome 14, analysis 2]

15. Secondary Outcome: Area Under the Curve (AUC) of Change From Baseline in Time to Culture Positivity in the MGIT System
Description: AUC of change from baseline for time to culture positivity (i.e., TTD) (Days 0 to 57), summarizes overall participant response for treatment period. Larger AUC of change from baseline for time to culture positivity would strongly suggest a clinical response with reduction of burden of MTB organisms in sputum. For this analysis, ti=visit day of each visit; t0=Day 0, t1=Day 8, t2=Day 15, etc. and xi=change from baseline in time to culture positivity at each visit; AUC at each visit was determined as AUCi=(ti - ti-1)(xi+ xi-1)/2. Average AUC of change from baseline was the sum of all AUCi divided by a given participant's duration in the trial up to 57 days. Baseline (Day 0)=the average of Day -1 and Day 1 values, if cultures on both days were positive; if only one culture was positive, value for time to culture positivity for positive culture was used as baseline.
Time Frame: Baseline to Day 57
Population: MITT Population included all participants who had sputum cultures positive for MDR TB at baseline (Day -1 and/or Day 1) using the MGIT system. Overall number analyzed are the participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 137 | 134 | 121
days | 13.4 (0.7) | 13.1 (0.7) | 11.1 (0.7)
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0246, ANCOVA; Pairwise comparison was derived from ANCOVA model with factors of treatment, baseline cavitation status and covariate baseline
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0529, ANCOVA; [statistical method as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Delamanid 100 mg BID + OBR vs Delamanid 200 mg BID + OBR; Test type: Superiority; p = 0.7508, ANCOVA; [statistical method as in outcome 15, analysis 1]

16. Secondary Outcome: Percentage of Participants With Sputum Culture Negative at Day 57 Using the MGIT System Without Consideration of Subsequent Culture Results
Time Frame: Day 57
Population: MITT Population included all participants who had sputum cultures positive for MDR TB at baseline (Day -1 and/or Day 1) using the MGIT system.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 141 | 136 | 125
percentage of participants | 56.0 | 52.9 | 44.0
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0518, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.272, 95% CI 2-sided [0.995 to 1.627]
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.1506, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.203, 95% CI 2-sided [0.934 to 1.550]

17. Secondary Outcome: Percentage of Participants With Sputum Culture Negative at Day 57 and Day 84 Using the MGIT System Without Respect to Interim Culture Results
Time Frame: Day 57 and Day 84
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 141 | 136 | 125
percentage of participants | 50.4 | 44.9 | 40.8
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.1201, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.234, 95% CI 2-sided [0.945 to 1.612]
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.5112, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.099, 95% CI 2-sided [0.829 to 1.456]

18. Secondary Outcome: Percentage of Participants With Sputum Culture Negative at Day 57 Using Solid Culture Media Without Respect to Subsequent Culture Results
Time Frame: Day 57
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 119 | 115 | 113
percentage of participants | 65.5 | 71.3 | 49.6
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0141, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.323, 95% CI 2-sided [1.053 to 1.661]
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.438, 95% CI 2-sided [1.155 to 1.791]

19. Secondary Outcome: Percentage of Participants With Sputum Culture Negative at Day 57 and Day 84 Using Solid Culture Media Without Respect to Interim Culture Results
Time Frame: Day 57 and Day 84
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 119 | 115 | 113
percentage of participants | 60.5 | 67.8 | 45.1
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0196, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.341, 95% CI 2-sided [1.044 to 1.722]
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; P-value was derived using CMH test stratified by randomization strata (cavitation); Risk Ratio Mean = 1.503, 95% CI 2-sided [1.183 to 1.909]

20. Secondary Outcome: Percentage of Participants Who Achieved SCC From the MGIT System Analyzed by Cochran-Armitage Linear Trend Test for Dose-response Relationship
Description: A participant achieving SCC using solid media is defined as one with sputum culture negative for growth of MTB on Day 57, and (a) not followed by a positive culture at any point thereafter, and (b) confirmed by at least one additional negative sputum culture at Day 84. A dose response in the percentage of participants achieving SCC using the MGIT system was tested by the Cochran-Armitage linear trend test with equally spaced dose scores (0, 1, and 2 for placebo, 100 mg BID, and 200 mg BID, respectively).
Time Frame: From the first dose of study drug up to the end of the Post-treatment Follow-up Period (Up to Day 84)
Population: MITT Population included all participants who had sputum cultures positive for multidrug resistant tuberculosis (MDR TB) at baseline (Day -1 and/or Day 1) using the MGIT system.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 141 | 136 | 125
percentage of participants | 45.4 | 41.9 | 29.6
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0468, Cochran-Armitage Linear Trend Test; Cochran-Armitage test was performed for dose response with the treatment group ordered as placebo, delamanid 100 mg BID, and delamanid 200 mg BID

21. Secondary Outcome: Percentage of Participants Who Achieved Initial SCC Using the MGIT System
Description: Initial SCC occurred at the time of the collection of the first sputum specimen with mycobacterial culture negative for growth of MTB using the MGIT system followed by at least one additional MGIT negative sputum specimen at least 27 days after the first negative specimen and no sputum specimens MGIT positive for growth at any point between the negative MGIT sputum specimens. Survival analysis methodology was performed to compare the Kaplan-Meier curves for time to SCC across 3 treatment groups. Comparisons between 100 mg BID and placebo and 200 mg BID and placebo were also performed with stratified log-rank tests. The benefit ratios (ratio of likelihoods that participants treated with delamanid BID + OBR would achieve SCC more rapidly than participants treated with placebo + OBR) for participants achieving SCC were computed.
Time Frame: Day 57
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 141 | 136 | 125
percentage of participants | 50.4 | 50.0 | 31.2
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0011, Stratified Log-Rank Test; p-value was derived from log-rank test with SAS Proc lifetest for comparisons with placebo; Hazard Ratio (HR) = 1.856, 95% CI 2-sided [1.255 to 2.745] — Hazard ratio computed with SAS PROC PHREG for comparisons with placebo
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0013, Stratified Log-Rank Test; p-value was derived from log-rank test with SAS Proc lifetest for comparisons with placebo; Hazard Ratio (HR) = 1.849, 95% CI 2-sided [1.246 to 2.743] — Hazard ratio computed with SAS PROC PHREG for comparisons with placebo

22. Secondary Outcome: Percentage of Participants Who Achieved Initial SCC Using the Solid Culture Media
Description: Initial SCC occurred at the time of the collection of the first sputum specimen with mycobacterial culture negative for growth of MTB using solid culture media that was followed by at least one additional negative sputum specimen at least 27 days after the first negative specimen and no sputum specimens positive for growth on solid culture media at any point between the negative sputum specimens using solid culture media. Survival analysis methodology was performed to compare the Kaplan-Meier curves for time to SCC across 3 treatment groups. Comparisons between 100 mg BID and placebo and 200 mg BID and placebo were also performed with stratified log-rank tests. The benefit ratios (ratio of likelihoods that participants treated with delamanid BID + OBR would achieve SCC more rapidly than participants treated with placebo + OBR) for participants achieving SCC were computed.
Time Frame: Day 57
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 119 | 115 | 113
percentage of participants | 60.5 | 68.7 | 37.2
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0004, Stratified Log-Rank Test; P-value was derived from Log-rank test with SAS PROC LIFETEST for comparisons with placebo; Hazard Ratio (HR) = 1.926, 95% CI 2-sided [1.315 to 2.820] — Hazard ratio computed with SAS PROC PHREG for comparisons with placebo
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p < .0001, Stratified Log-Rank Test; Hazard Ratio (HR) = 2.190, 95% CI 2-sided [1.504 to 3.189]

23. Secondary Outcome: Percentage of Participants Who Achieved Final SCC Using MGIT
Description: Final SCC was defined as SCC at Day 57 or the latest time point of the first negative sputum culture establishing SCC for a given participant after the last positive sputum culture observed during the 56-day treatment period, whichever comes first. Survival analysis methodology was performed to compare the Kaplan-Meier curves for time to SCC across 3 treatment groups. Comparisons between 100 mg BID and placebo and 200 mg BID and placebo were also performed with stratified log-rank tests. The benefit ratios (ratio of likelihoods that participants treated with delamanid BID + OBR would achieve SCC more rapidly than participants treated with placebo + OBR) for participants achieving SCC were computed.
Time Frame: Day 57
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 141 | 136 | 125
percentage of participants | 45.4 | 41.9 | 29.6
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0056, Stratified Log-Rank Test; P-value was derived from Log-rank test with SAS PROC LIFETEST for comparisons with placebo; Hazard Ratio (HR) = 1.727, 95% CI 2-sided [1.152 to 2.591] — Hazard ratio computed with SAS PROC PHREG for comparisons with placebo
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0232, Stratified Log-Rank Test; P-value was derived from Log-rank test with SAS PROC LIFETEST for comparisons with placebo; Hazard Ratio (HR) = 1.585, 95% CI 2-sided [1.048 to 2.399] — Hazard ratio computed with SAS PROC PHREG for comparisons with placebo

24. Secondary Outcome: Percentage of Participants Who Achieved Final SCC Using Solid Culture Media
Description: Final SCC is defined as SCC at Day 57 or the latest time point of the first negative sputum culture establishing SCC for a given participant after the last positive sputum culture observed during the 56-day treatment period, whichever comes first. Survival analysis methodology was performed to compare the Kaplan-Meier curves for time to SCC across 3 treatment groups. Comparisons between 100 mg BID and placebo and 200 mg BID and placebo were also performed with stratified log-rank tests. The benefit ratios (ratio of likelihoods that participants treated with delamanid BID + OBR would achieve SCC more rapidly than participants treated with placebo + OBR) for participants achieving SCC were computed.
Time Frame: Day 57
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 119 | 115 | 113
percentage of participants | 53.8 | 65.2 | 33.6
Statistical Analysis 1: Comparison: Delamanid 100 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p = 0.0016, Stratified Log-Rank Test; P-value was derived from log-rank test with SAS PROC LIFETEST for comparisons with placebo; Hazard Ratio (HR) = 1.846, 95% CI 2-sided [1.235 to 2.759] — Hazard ratio computed with SAS PROC PHREG for comparisons with placebo
Statistical Analysis 2: Comparison: Delamanid 200 mg BID + OBR vs Placebo + OBR; Test type: Superiority; p < .0001, Stratified Log-Rank Test; P-value was derived from Log-rank test with SAS PROC LIFETEST for comparisons with placebo; Hazard Ratio (HR) = 2.301, 95% CI 2-sided [1.555 to 3.405] — Hazard ratio computed with SAS PROC PHREG for comparisons with placebo

25. Secondary Outcome: Percentage of Participants With Clinically Significant Physical Examination Findings, Including Vision and Neuropsychiatric Assessments
Time Frame: From first dose of study drug up to post treatment period (Day 84)
Population: ITT population included all randomized participants who received any amount of IMP, regardless of any protocol deviation or violation.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants | 0 | 0 | 0

26. Secondary Outcome: Percentage of Participants With Clinically Significant Vital Sign Abnormalities
Description: Criteria for potentially clinically significant vital sign abnormalities: Heart rate [beats per minute (BPM)]: >=120, increase >=15, <=60, decrease >=15; systolic blood pressure [millimeter of mercury (mmHg)]: >=160, increase >=20, <=90, decrease >=20; diastolic blood pressure (mmHg): >=105, increase >=15, <=50, decrease >=15; weight (kg) gain: increase >=5%; or weight loss: decrease >=5%; temperature [degrees Celsius (C)]: >=38.5, increase of >=1.1. Only categories with at least 1 participant with event are reported.
Time Frame: From first dose of study drug up to post treatment period (Day 84)
Population: ITT population included all randomized participants who received any amount of IMP, regardless of any protocol deviation or violation. Number analyzed is the number of participants who had at least one post-baseline numerical result for the given test.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants
  Weight: Decrease of >=5% in Body Weight: number analyzed (Participants) | 159 | 158 | 157
  Weight: Decrease of >=5% in Body Weight | 16.4 | 13.9 | 6.4
  Weight: Increase of >=5% in Body Weight: number analyzed (Participants) | 159 | 158 | 157
  Weight: Increase of >=5% in Body Weight | 35.2 | 32.3 | 44.6
  Temperature: >=38.5C + Increase of >=1.1C: number analyzed (Participants) | 159 | 158 | 157
  Temperature: >=38.5C + Increase of >=1.1C | 0.0 | 0.6 | 0.0
  Heart Rate: <=60 BPM + Decrease of >=15: number analyzed (Participants) | 159 | 158 | 158
  Heart Rate: <=60 BPM + Decrease of >=15 | 4.4 | 5.1 | 2.5
  Heart Rate: >=120 BPM + Increase of >=15: number analyzed (Participants) | 159 | 158 | 158
  Heart Rate: >=120 BPM + Increase of >=15 | 0.6 | 0.6 | 0.0
  Systolic Blood Pressure: <=90 mmHg + Decrease of >=20 mmHg: number analyzed (Participants) | 159 | 158 | 158
  Systolic Blood Pressure: <=90 mmHg + Decrease of >=20 mmHg | 4.4 | 9.5 | 8.9
  Systolic Blood Pressure: >=160 mmHg + Increase of >=20 mmHg: number analyzed (Participants) | 159 | 158 | 158
  Systolic Blood Pressure: >=160 mmHg + Increase of >=20 mmHg | 0.6 | 0.0 | 0.0
  Diastolic Blood Pressure <=50 mmHg + Decrease of >=15 mmHg: number analyzed (Participants) | 159 | 158 | 158
  Diastolic Blood Pressure <=50 mmHg + Decrease of >=15 mmHg | 1.9 | 0.0 | 0.6

27. Secondary Outcome: Percentage of Participants With Categorical Changes in 12-lead Electrocardiogram Results at Day 56
Description: Criteria for categorical changes in 6 12-lead Electrocardiogram results: Vent Rate Outliers Notable Decreases- >= 25% decrease from Baseline and ventricular rate < 50 beats per minute (beats/min), notable increases- >= 25% decrease from Baseline and ventricular rate > 100 beats/min; PR outliers notable changes- >= 25% change from Baseline when PR > 200 milliseconds (msec); QRS outliers notable changes- >= 25% change from Baseline when QRS > 100 msec; QT new onset (> 500 msec); QT correction with Bazett formula (QTcB) and QT interval with Fridericia's correction (QTcF) new onset > 500 msec, > 480 msec, > 450 msec, where new onset (> 450, 480, 500 msec) means a participant who attains a value > 450, 480, 500 msec during Treatment Period but not at each Baseline Visit; change >= 30, <= 60 msec; change > 60 msec; and new abnormal U waves, ST segment changes, T wave changes, abnormal rhythm, RBBB, LBBB, myocardial infarction(MI). Only categories with at least 1 participant with event are r
Time Frame: Baseline up to Day 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants
  Vent Rate Outliers Notable Decreases | 0.0 | 1.2 | 0.6
  Vent Rate Outliers Notable Increases | 1.2 | 2.5 | 3.7
  QT New Onset (> 500 msec) | 0.0 | 1.8 | 0.0
  QTcB New Onset (> 500 msec) | 1.2 | 1.2 | 1.2
  QTcB New Onset (> 480 msec) | 7.4 | 8.1 | 3.1
  QTcB New Onset (> 450 msec) | 39.1 | 37.5 | 19.3
  QTcB Change >= 30, <= 60 msec | 36.6 | 44.3 | 17.5
  QTcB Change >60 msec | 1.2 | 3.1 | 0.6
  QTcF New Onset (> 480 msec) | 0.0 | 3.1 | 0.6
  QTcF New Onset (> 450 msec) | 15.5 | 13.7 | 6.2
  QTcF Change >= 30, <= 60 msec | 36.0 | 44.3 | 15.6
  QTcF Change > 60 msec | 3.1 | 3.7 | 0.0
  New Abnormal Rhythm | 9.3 | 10.6 | 17.5
  New Right Bundle Branch Block (RBBB), Left Bundle Branch Block (LBBB), Myocardial Infarction (MI) | 2.4 | 3.7 | 7.5

28. Secondary Outcome: Percentage of Participants With Clinically Significant Laboratory Test Abnormalities
Description: The laboratory values were one of the parameters to measure the safety and tolerability of individual participants. Participants with potentially clinically significant laboratory values in clinical chemistry, hematology, coagulation, adrenal function tests, urinalysis and thyroid function tests that were identified based on pre-defined criteria were reported. Any value outside the normal range was flagged for the attention of the investigator who assessed whether or not a flagged value is of clinical significance. The categories with at least one participant with abnormal lab value as assessed by the investigator are reported.
Time Frame: From first dose of study drug up to post treatment period (Day 84)
Population: ITT population included all randomized participants who received any amount of IMP, regardless of any protocol deviation or violation. Number analyzed is the number of participants with at least one non-missing result for a given lab test.
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants
  Albumin (grams per deciliter [g/dL]) <2.6 | 8.1 | 3.1 | 8.8
  Alanine Transaminase (ALT) (units per liter [U/L]) >150.0 | 0.6 | 0.6 | 1.3
  Aspartate aminotransferase (AST) (U/L) >150.0 | 1.2 | 1.9 | 2.5
  Bilirubin, Total (mg/dL) >2: number analyzed (Participants) | 0 | 160 | 0
  Bilirubin, Total (mg/dL) >2 |  | 0.6 |
  Calcium (mg/dL) <7, >11.5: number analyzed (Participants) | 160 | 159 | 160
  Calcium (mg/dL) <7, >11.5 | 0.6 | 1.9 | 3.8
  Chloride (milliequivalents per liter [mEq/L]) <85 | 0.6 | 2.5 | 0.6
  Cholesterol (mg/dL) >300.0: number analyzed (Participants) | 161 | 160 | 0
  Cholesterol (mg/dL) >300.0 | 0.6 | 0.6 |
  Creatinine (mg/dL) >2.0 | 1.2 | 0.6 | 1.9
  Gamma-glutamyl Transferase (U/L); Male >225.0, Female >175.0: number analyzed (Participants) | 161 | 0 | 160
  Gamma-glutamyl Transferase (U/L); Male >225.0, Female >175.0 | 3.1 |  | 1.3
  Glucose (mg/dL) <50, >300 | 1.9 | 1.9 | 4.4
  Lactic Dehydrogenase (U/L) >400 | 1.2 | 3.8 | 1.9
  Potassium (mEq/L) <3, >5.5 | 16.1 | 18.1 | 18.1
  Protein, Total Serum (g/dL) >9.5: number analyzed (Participants) | 161 | 0 | 0
  Protein, Total Serum (g/dL) >9.5 | 0.6 |  |
  Sodium (mEq/L) <132, >148 | 17.4 | 16.3 | 17.5
  Triglycerides (mg/dL) >300 | 4.3 | 3.8 | 4.4
  Urea Nitrogen (mg/dL) >34 | 1.9 | 1.3 | 1.9
  Uric Acid (mg/dL) >12: number analyzed (Participants) | 153 | 154 | 157
  Uric Acid (mg/dL) >12 | 24.2 | 27.9 | 22.9
  Activated Partial Thromboplastin Time (seconds [sec]) >45.0 | 14.9 | 12.5 | 16.3
  Eosinophils, Absolute (thousands per microliter [thous/µL]) >=0.8 | 14.9 | 18.1 | 24.4
  Hematocrit (%); Male <32, >58, Female <27, >58 | 15.5 | 11.3 | 11.3
  Hemoglobin (g/dL) <10, >16 | 28.6 | 23.1 | 22.5
  Lymphocytes, Absolute (thous/µL) >=5.0: number analyzed (Participants) | 161 | 0 | 160
  Lymphocytes, Absolute (thous/µL) >=5.0 | 0.6 |  | 1.3
  Mean Corpuscular Hemoglobin (picograms [pg]) >40.0: number analyzed (Participants) | 161 | 0 | 0
  Mean Corpuscular Hemoglobin (picograms [pg]) >40.0 | 0.6 |  |
  Mean Corpuscular Hemoglobin Concentrate (g/dL) >40.0: number analyzed (Participants) | 0 | 0 | 160
  Mean Corpuscular Hemoglobin Concentrate (g/dL) >40.0 |  |  | 0.6
  Mean Corpuscular Volume (femtoliter [fL]) <=78, >=105 | 30.4 | 26.3 | 26.9
  Neutrophil, Bands (%) >=8.0: number analyzed (Participants) | 76 | 77 | 78
  Neutrophil, Bands (%) >=8.0 | 2.6 | 2.6 | 1.3
  Neutrophils, Absolute (thous/µL) <=2.0 | 13.7 | 10.0 | 13.8
  Platelet Count (thous/µL) <100, >600 | 16.1 | 15.6 | 13.8
  Prothrombin Time (sec) >17.5: number analyzed (Participants) | 129 | 134 | 138
  Prothrombin Time (sec) >17.5 | 4.7 | 3.7 | 1.4
  Red Blood Cell (RBC) Count (million per microliter [mill/µL]) <4, >=6.5 | 31.7 | 23.1 | 26.3
  Reticulocyte Count (%) <=.1, >=3 | 21.1 | 21.3 | 23.8
  White Blood Count (thous/µL) <3, >=15 | 11.2 | 12.5 | 13.8
  Blood (Urinalysis): Positive: number analyzed (Participants) | 156 | 157 | 157
  Blood (Urinalysis): Positive | 55.8 | 58.6 | 55.4
  Epithelial Casts: number analyzed (Participants) | 4 | 9 | 5
  Epithelial Casts | 100.0 | 100.0 | 100.0
  Granular Cast: number analyzed (Participants) | 11 | 8 | 6
  Granular Cast | 100.0 | 100.0 | 100.0
  Hyaline Cast: number analyzed (Participants) | 17 | 10 | 12
  Hyaline Cast | 100.0 | 100.0 | 100.0
  RBC Casts: number analyzed (Participants) | 0 | 1 | 1
  RBC Casts |  | 100.0 | 100.0
  White Blood Count Casts: number analyzed (Participants) | 2 | 2 | 0
  White Blood Count Casts | 100.0 | 100.0 |
  Cortisol, Serum (micrograms per deciliter [µg/dL]) >=26 | 36.0 | 48.8 | 29.4
  Free Thyroxine (T4) [nanograms per deciliter (ng/dL)] <=.30, >=2.5: number analyzed (Participants) | 157 | 156 | 156
  Free Thyroxine (T4) [nanograms per deciliter (ng/dL)] <=.30, >=2.5 | 1.9 | 0.6 | 1.3
  Thyroid Stimulating Hormone (micro-international units per milliliter [µIU/mL]) <=.30 >=3: number analyzed (Participants) | 157 | 155 | 156
  Thyroid Stimulating Hormone (micro-international units per milliliter [µIU/mL]) <=.30 >=3 | 23.6 | 20.0 | 26.3

29. Secondary Outcome: Percentage of Participants With Clinically Significant Audiometry Findings
Time Frame: From first dose of study drug up to post treatment period (Day 84)
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants | 0 | 0 | 0

30. Secondary Outcome: Percentage of Participants Using Concomitant Medications
Description: The concomitant anti-TB medication were classified as per WHO 2008 guidelines and included: Category 1- first-line oral anti-tuberculosis drugs; Category 2- injectable anti-tuberculosis drugs; Category 3- fluoroquinolones; Category 4- oral bacteriostatic second-line anti-tuberculosis drugs; Category 5- anti-tuberculosis drugs with unclear efficacy or unclear role in MDR-TB treatment (not recommended by WHO for routine use in MDR-TB participants).
Time Frame: From first dose of study drug up to post treatment period (Day 84)
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants
  Concomitant Medications (Excluding Anti-TB Medications) | 98.8 | 98.8 | 98.8
  Concomitant Anti-TB Medications: Category 1 | 90.7 | 90.6 | 88.8
  Concomitant Anti-TB Medications: Category 2 | 88.2 | 80.0 | 88.8
  Concomitant Anti-TB Medications: Category 3 | 97.5 | 98.8 | 98.1
  Concomitant Anti-TB Medications: Category 4 | 99.4 | 98.8 | 99.4
  Concomitant Anti-TB Medications: Category 5 | 26.1 | 27.5 | 27.5

31. Secondary Outcome: Percentage of Participants With At Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical trial participant and which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including e.g., an abnormal laboratory assessment result), symptom or disease temporally associated with participation in the clinical trial, whether or not it is considered causally related to the medicinal product or procedures of the clinical trial. A clinically significant worsening in the health of the participant compared with the participant's health status documented at baseline constituted a TEAE.
Time Frame: From first dose of study drug up to post treatment period (Day 84)
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants | 90.1 | 93.1 | 93.1

32. Secondary Outcome: Time-matched Change From Baseline (Day -1) in QTcF at Day 56
Time Frame: Baseline, and 2, 3, 4, 10, 12, and 24 hours post dose on Day 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
msec
  Day 56: 2 Hours Post Dose | 11.8 (16.3) | 14.6 (18.8) | -0.5 (14.3)
  Day 56: 3 Hours Post Dose | 12.8 (16.6) | 14.7 (16.0) | -0.4 (14.5)
  Day 56: 4 Hours Post Dose | 16.8 (16.3) | 19.4 (17.3) | 5.0 (15.8)
  Day 56: 10 Hours Post Dose | 16.5 (17.4) | 20.8 (17.3) | 5.2 (15.5)
  Day 56: 12 Hours Post Dose | 15.6 (17.4) | 16.7 (17.0) | 2.6 (15.6)
  Day 56: 24 Hours Post Dose | 15.5 (18.9) | 18.3 (18.5) | 3.4 (15.0)

33. Secondary Outcome: Mean Change From Baseline in QTcF
Time Frame: Baseline, Days 1, 14, 28 and 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
msec
  Day 1 | 0.1 (7.1) | 0.0 (7.1) | -1.8 (8.3)
  Day 14 | 7.7 (11.1) | 9.3 (11.2) | 0.8 (11.0)
  Day 28 | 9.9 (12.3) | 14.1 (13.2) | 2.4 (11.2)
  Day 56 | 14.9 (14.3) | 17.5 (13.9) | 2.7 (12.2)

34. Secondary Outcome: Mean Change From Baseline in QTcB
Time Frame: Baseline, Days 1, 14, 28 and 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
msec
  Day 1 | 0.8 (7.4) | 1.5 (7.2) | -0.4 (8.5)
  Day 14 | 6.5 (11.5) | 8.1 (10.7) | 0.5 (12.0)
  Day 28 | 7.9 (12.1) | 12.5 (14.0) | 2.1 (13.0)
  Day 56 | 11.7 (14.5) | 14.6 (12.6) | 2.3 (13.6)

35. Secondary Outcome: Mean Change From Baseline in Ventricular Rate
Time Frame: Baseline, Days 1, 14, 28 and 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
beats/min
  Day 1 | 0.9 (5.5) | 2.0 (4.9) | 1.9 (5.3)
  Day 14 | -1.9 (8.1) | -2.1 (9.0) | -0.6 (8.6)
  Day 28 | -3.2 (8.6) | -3.2 (9.3) | -0.8 (10.2)
  Day 56 | -4.8 (10.3) | -4.7 (12.6) | -1.2 (10.6)

36. Secondary Outcome: Mean Change From Baseline in PR Interval
Time Frame: Baseline, Days 1, 14, 28 and 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
msec
  Day 1 | -1.3 (5.6) | -1.0 (4.8) | -1.6 (5.4)
  Day 14 | -0.7 (7.7) | -0.8 (7.2) | -1.4 (8.1)
  Day 28 | -1.4 (8.1) | -0.8 (8.4) | -0.6 (7.4)
  Day 56 | -1.6 (8.3) | 0.3 (8.1) | -0.5 (7.2)

37. Secondary Outcome: Mean Change From Baseline in QRS Interval
Time Frame: Baseline, Days 1, 14, 28 and 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
msec
  Day 1 | -0.3 (2.8) | -0.5 (2.8) | -0.2 (3.3)
  Day 14 | 0.1 (3.3) | 0.1 (3.5) | -0.1 (3.9)
  Day 28 | 0.4 (3.6) | -0.1 (4.2) | -0.3 (3.8)
  Day 56 | 0.7 (4.1) | -0.2 (4.0) | 0.2 (3.8)

38. Secondary Outcome: Mean Change From Baseline in QT Interval
Time Frame: Baseline, Days 1, 14, 28 and 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
msec
  Day 1 | -1.0 (11.5) | -2.7 (10.9) | -4.3 (11.6)
  Day 14 | 9.5 (18.2) | 11.1 (20.1) | 1.1 (18.5)
  Day 28 | 13.4 (20.3) | 16.3 (21.1) | 2.5 (20.2)
  Day 56 | 20.1 (23.5) | 22.0 (28.4) | 3.1 (21.7)

39. Secondary Outcome: Percentage of Participants With Change in ECG Morphological Patterns From Baseline
Description: Any changes in the ECG waves or segments as assessed by the investigator were reported.
Time Frame: Baseline, Days 1, 14, 28 and 56
Population: The ECG population included all participants who had at least one baseline and one on-treatment ECG (full data set).
Measure: Number; unit: percentage of participants
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
Number analyzed (Participants) | 161 | 160 | 160
percentage of participants
  Day 1: New Abnormal U Waves | 0.0 | 0.0 | 0.0
  Day 1: New ST Segment Changes | 1.8 | 0.6 | 1.2
  Day 1: New T Wave Changes | 9.9 | 6.2 | 6.2
  Day 14: New Abnormal U Waves | 0.0 | 0.0 | 0.0
  Day 14: New ST Segment Changes | 3.1 | 0.6 | 1.2
  Day 14: New T Wave Changes | 12.4 | 5.6 | 4.3
  Day 28: New Abnormal U Waves | 1.2 | 0.0 | 0.0
  Day 28: New ST Segment Changes | 1.8 | 0.0 | 0.0
  Day 28: New T Wave Changes | 11.8 | 5.0 | 10.0
  Day 56: New Abnormal U Waves | 1.2 | 0.6 | 0.0
  Day 56: New ST Segment Changes | 2.4 | 0.6 | 1.8
  Day 56: New T Wave Changes | 11.1 | 10.6 | 5.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to post treatment period (up to Day 84)
Description: ITT population included all randomized participants who received any amount of IMP, regardless of any protocol deviation or violation.
Arm/Group | Delamanid 100 mg BID + OBR | Delamanid 200 mg BID + OBR | Placebo + OBR
All-Cause Mortality (participants affected / at risk) | 0/161 | 1/160 | 0/160
Serious Adverse Events (participants affected / at risk) | 16/161 | 20/160 | 14/160
Other Adverse Events (participants affected / at risk) | 145/161 | 148/160 | 147/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid 100 mg BID + OBR (N=161) | Delamanid 200 mg BID + OBR (N=160) | Placebo + OBR (N=160)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 7 | 9 | 3
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Agitation (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Delusional disorder, persecutory type (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0
Ideas of reference (Psychiatric disorders) | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 2 | 3
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delamanid 100 mg BID + OBR (N=161) | Delamanid 200 mg BID + OBR (N=160) | Placebo + OBR (N=160)
Anaemia (Blood and lymphatic system disorders) | 15 | 8 | 14
Eosinophilia (Blood and lymphatic system disorders) | 7 | 11 | 15
Reticulocytosis (Blood and lymphatic system disorders) | 19 | 20 | 17
Palpitations (Cardiac disorders) | 13 | 20 | 10
Tinnitus (Ear and labyrinth disorders) | 16 | 22 | 12
Vision blurred (Eye disorders) | 12 | 15 | 9
Abdominal discomfort (Gastrointestinal disorders) | 7 | 8 | 5
Abdominal distension (Gastrointestinal disorders) | 5 | 9 | 5
Abdominal pain (Gastrointestinal disorders) | 16 | 12 | 11
Abdominal pain lower (Gastrointestinal disorders) | 4 | 11 | 7
Abdominal pain upper (Gastrointestinal disorders) | 41 | 36 | 38
Constipation (Gastrointestinal disorders) | 6 | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 20 | 12 | 22
Dyspepsia (Gastrointestinal disorders) | 6 | 14 | 6
Gastritis (Gastrointestinal disorders) | 8 | 14 | 16
Nausea (Gastrointestinal disorders) | 58 | 65 | 53
Toothache (Gastrointestinal disorders) | 6 | 7 | 11
Vomiting (Gastrointestinal disorders) | 48 | 58 | 44
Asthenia (General disorders) | 20 | 27 | 20
Chest pain (General disorders) | 16 | 13 | 7
Injection site pain (General disorders) | 13 | 12 | 23
Malaise (General disorders) | 12 | 16 | 12
Pyrexia (General disorders) | 9 | 18 | 18
Electrocardiogram QT prolonged (Investigations) | 11 | 13 | 3
Anorexia (Metabolism and nutrition disorders) | 23 | 34 | 24
Hyperuricaemia (Metabolism and nutrition disorders) | 31 | 38 | 35
Hypokalaemia (Metabolism and nutrition disorders) | 20 | 29 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 43 | 46
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 16 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 8 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 21 | 26
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 8 | 8
Dizziness (Nervous system disorders) | 48 | 49 | 49
Dysgeusia (Nervous system disorders) | 5 | 10 | 10
Headache (Nervous system disorders) | 36 | 41 | 30
Hypoaesthesia (Nervous system disorders) | 12 | 7 | 8
Paraesthesia (Nervous system disorders) | 17 | 20 | 12
Somnolence (Nervous system disorders) | 11 | 9 | 15
Tremor (Nervous system disorders) | 19 | 16 | 13
Anxiety (Psychiatric disorders) | 9 | 11 | 5
Depression (Psychiatric disorders) | 4 | 13 | 5
Insomnia (Psychiatric disorders) | 42 | 51 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 16 | 14 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 6
Rales (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 16
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 17 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 15 | 20
Rash (Skin and subcutaneous tissue disorders) | 8 | 3 | 10
Rash papular (Skin and subcutaneous tissue disorders) | 10 | 12 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.